CLINICAL TRIAL: NCT06848933
Title: Could the Advanced Hybrid Closed-Loop System Algorithm Provide Postprandial Normoglycemia After a High-Fat, High-Protein Meal
Acronym: AHCLS T1D nutr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Izmir Tinaztepe University (Other)
Responsible Party: Principal Investigator, Yasemin Atik Altinok, Dietician, PhD, Assoc Prof, Izmir Tinaztepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AHCLS T1D high fat and protein
Record Dates: First submitted 2024-11-28; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes Mellitus; Adolescents
Keywords: AHCLS; type 1 diabetes; high fat, high protein; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Adolescents with type 1 diabetes on Medtronic Minimed 780G (Experimental): Each participant will consume the test meal in Medtronic Minimed 780Gmanual mode and Medtronic Minimed 780G in auto mode. Each participant will be in control of himself/herself
  Interventions: Other: Test meal; Device: Each participant will consume the test meal when on Medtronic Minimed 780G and will consume test meal on Medtronic Minimed 780G on manual mode; Device: Advanced hybrid closed loop system mode

INTERVENTIONS:
Other: Test meal — On days 1, 2 and 3 of the study, a pediatric endocrinologist from the research team will evaluate the continuous glucose monitoring system data and optimize the carbohydrate/insulin ratios. On days 4 and 7 of the study, participants with blood sugar levels between 70-140 mg/dl according to the continuous glucose monitoring system, which is a component of the hybrid closed-loop insulin infusion pump system, will consume the test meal consisting of Dr Oetker Ristorante Pizza Mista (340 grams) (92 g carbohydrate, 33 g protein, 41 g fat) at lunch, under the supervision of a dietician from the research team, by switching the pump to manual mode and entering the carbohydrate amount of the meal into the pump. This application will be repeated on days 11 and 14 of the study, with the participant's pump in automatic mode. Participants will not be allowed to consume food or beverages other than water or exercise for 5 hours after the meal. Blood sugar monitoring will be done with the continuous
Device: Each participant will consume the test meal when on Medtronic Minimed 780G and will consume test meal on Medtronic Minimed 780G on manual mode — After the intervention, blood glucose values will be documented from continued glucose measurement system for postprandial 5 hours,and compared in manual mode and auto mode
Device: Advanced hybrid closed loop system mode — On days 1, 2 and 3 of the study, a pediatric endocrinologist from the research team will evaluate the continuous glucose monitoring system data and optimize the carbohydrate/insulin ratios. On days 4 and 7 of the study, participants with blood sugar levels between 70-140 mg/dl according to the continuous glucose monitoring system, which is a component of the hybrid closed-loop insulin infusion pump system, will consume the test meal consisting of Dr Oetker Ristorante Pizza Mista (340 grams) (92 g carbohydrate, 33 g protein, 41 g fat) at lunch, under the supervision of a dietician from the research team, by switching the pump to manual mode and entering the carbohydrate amount of the meal into the pump. This application will be repeated on days 11 and 14 of the study, with the participant's pump in automatic mode. Participants will not be allowed to consume food or beverages other than water or exercise for 5 hours after the meal. Blood sugar monitoring will be done with the continuous

SUMMARY:
AHCL Systems Could Cover Postprandial Glycemic Response After High Fat and High Protein Meals

DETAILED DESCRIPTION:
On the 1st, 2nd and 3rd day of the study, a pediatric endocrinologist from the research team will evaluate the continuous glucose measurement system data and optimize the carbohydrate/insulin ratios. On the 4th and 7th days of the study, participants with blood sugar levels between 70-140 mg/dl according to the continuous glucose measurement system, which is a component of the hybrid closed-loop insulin infusion pump system, will consume the test meal consisting of Dr Oetker Ristorante Pizza Mista (340 grams) (92 g carbohydrate, 33 g protein, 41 g fat) at lunch, under the supervision of a dietician from the research team, by switching the pump to manual mode and entering the carbohydrate amount of the meal into the pump. This application will be repeated on the 11th and 14th days of the study while the participant's pump is in automatic mode. Participants will not be allowed to consume food or beverages other than water or exercise for 5 hours after the meal. Blood sugar monitoring will be done with a continuous glucose measurement system. The participant will leave the hospital 5 hours after the start of the meal to return to their normal life. Dr Oetker Ristorante Pizza Mista, which was selected as the test meal, was chosen because it is a macronutrient content that is consumed by young people between the ages of 9-18 and that is similar to the test meals in the world literature and accepted research reports reporting the effect of high-fat and high-protein meals on glycemic response in individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Not having a disease accompanying type 1 diabetes (celiac, cystic fibrosis, etc.)

Exclusion Criteria:

* - Not volunteering to participate in the study
* Using psychiatric medication or any medication that may cause obesity at the time of trial
* Having a disease accompanying type 1 diabetes (celiac, cystic fibrosis, etc.)

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
time spend in time in range (70-180 mg/dl) for postprandial 5 hours after the test meal | 1 month
  Percentage of time when blood sugar is at 70-180 mg/dl for pst prandial 5 hours after the test meal

CONTACTS AND LOCATIONS:
Overall Officials: yasemin atik altınok, Assoc Prof, Principal Investigator — İzmir Tınaztepe University; Damla Goksen, Prof Dr, Study Director — Ege University
Locations (1):
- Ege University, Medical Faculty, Division of Pediatric Endocrinology, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided